CLINICAL TRIAL: NCT01324245
Title: Paracrine Regulation of Renal Function by Dopamine in Normotensive Humans
Brief Title: Intervention Study to Compare the Natriuretic Effects of Enalapril on Low and High Salt Diet
Acronym: Salt
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Georgetown University (Other)
Collaborators: University of Virginia (Other)
Responsible Party: Aruna R Natarajan/ Assistant Professor, Georgetown University Hospital
Allocation: Randomized | Model: Crossover | Masking: Quadruple
Other Study IDs: 2003-142; RR 17613 (Other: National Center for Research resources, NIH)
Record Dates: First submitted 2011-03-25; First posted 2011-03-28 (Estimated); Last update posted 2011-03-28 (Estimated); Status verified 2003-11

CONDITIONS: Salt-sensitive Hypertension
Keywords: Salt; Balance; Renin Angiotensin System; Fenoldopam\blood Pressure; Sodium
MeSH Terms: interventions — Fenoldopam; Enalaprilat

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Enalapril (Experimental): 2.5 mg every 12 hours for two doses
  Interventions: Drug: Fenoldopam

INTERVENTIONS:
Drug: Fenoldopam — Intravenous infusion at 0.5 mics/Kg/min for three hours
  Other Names: Enalaprilat; Corlopam

SUMMARY:
The kidney plays a crucial role in maintaining salt balance by two opposing physiological mechanisms: the renal dopaminergic system which enhances salt excretion and the renin-angiotensin system (RAS) which causes salt retention. Salt-sensitive hypertension occurs when this balance is altered or abnormal. We hypothesized that this balance is influenced by salt intake: therefore dietary salt affects the natriuretic response to the renal dopaminergic agonist Fenoldopam, and the Angiotensin Converting Enzyme inhibitor, Enalapril.

In this trial we study normal salt balance mechanisms in salt resistant adults with normal blood pressure.

DETAILED DESCRIPTION:
Eight adults of both genders and all races were studied in this double blind placebo controlled cross over study with randomization of the order of interventions. After 5 days each on low salt (about 1 gram/day) and high salt (about 6 grams/day)diet, with a washout period of at least four weeks in between, every subject was treated with Enalapril and Placebo on two consecutive days, followed by a Fenoldopam infusion for three hours, during which natriuresis and renal function testing were performed.

ELIGIBILITY:
Inclusion Criteria:

* Volunteers
* Healthy
* Normal Blood Pressure

Exclusion Criteria:

* Renal Impairment
* Obesity
* Salt sensitive increase in blood pressure

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 45 (Actual)
Dates: Start 2002-11; Primary Completion 2005-12 (Actual); Study Completion 2006-05 (Actual)

PRIMARY OUTCOMES:
Urinary sodium excretion | During the trial: a 3 hour fenoldopam infusion
  All subjects received placebo/enalapril in a randomized counterbalanced fashion in both phases. Phase 1 was on low salt, while Phase 2 was on high salt. All subjects received a 3 hour fenoldopam infusion, during which time urinary sodium excretion was measured as the primary outcome bvariable.

SECONDARY OUTCOMES:
Renal Plasma Flow | During 3 hour fenoldopam infusion
  In order to explain physiologically the effects of fenoldopam on urinary sodium excretion on high and low salt diet, with and wothout enalapril, renal plasma flow was measured during the infusion using PAH clearance

CONTACTS AND LOCATIONS:
Overall Officials: Aruna R Natarajan, MD, PhD, Principal Investigator — Georgetown University Hospital; Pedro A Jose, MD, PhD, Study Director — Georgetown University/ George Washington University
Locations (1):
- Georgetown University Medical Center, Washington D.C., District of Columbia, United States